CLINICAL TRIAL: NCT02581098
Title: Novel Regulators of Wound Angiogenesis and Inflammation
Brief Title: miR-200b & miR-21 in Diabetic Wounds
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Chandan Sen, Professor, Indiana University
Other Study IDs: 1807426080; GM108014/DK114718 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Foot Ulcer; Ulcer; Diabetic Foot Ulcer; Wound; Wound Heal
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Ulcer; Diabetic Foot; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, wound fluid
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
This study aims to determine if elevated wound-edge endothelial miR-200b is a barrier to wound healing in diabetic patients and also to determine if ex vivo supplementation of miR-21 mimic and recombinant MFG-E8 resolve inflammation in wound macrophages isolated from NPWT sponges from diabetic wounds. This study will enroll 124 (60 in the miR-200b arm and 64 in the miR21 arm) Diabetic Wound patients who have wound tissue oxygenation adequate to support wound healing and will be in the study for 14 weeks that includes 4 study visits.

DETAILED DESCRIPTION:
The study is designed as a 14 week prospective observational study where patients with diabetic wounds visiting the Indiana University Health Comprehensive Wound Center (CWC) will be enrolled. Patients enrolled will be followed for 14 weeks including 4 study visits, initial visit (week 0), study visit 2 (week 2), study visit 3 (week 4), and will return for a final follow-up study visit 4 (week 14; miR-200b arm only). Standardized Care Outline will be per physician discretion.

The initial visit will take place during the patients regularly scheduled CWC visit and the following will take place: informed consent will be obtained, baseline demographics and medical history with be collected, current labs and medications will be recorded, wound data will be obtained, an ankle brachial index will be completed for patients with leg wounds below the knee, if not already completed per Standard of Care (SoC) since onset of the wound, and wound photographs for digital planimetry to measure wound area. Wound fluid will be collected using a filter paper method, aspiration method, or via the NPWT (Negative Pressure Wound Therapy, also known as Wound Vac) sponge prior to debridement. Additionally, two 3 mm punch tissue biopsies will be obtained from the patient's physician; however, this is optional. If the wound shows signs of healing and does not show signs of infection (i.e. the wound has not stalled in healing for 2 or more weeks or become larger in size) or the wound has been declared healed by their physician, the biopsies will not be obtained. The study visits 2-4 will include the following: a medication and adverse event review, wound data will be recorded, wound photographs, wound fluid, and two 3 mm punch tissue biopsies will be obtained from the patient's physician.

Potential Risks:

The risks associated with this research study are low. There are no therapeutic interventions or medications as part of this study to be administered depending on the amount of sensation the subject has at the site of the wound.

If the subject is receiving a biopsy, the wound site will be numbed by applying local anesthesia as appropriate to the area being biopsied. There may be some discomfort with the tissue biopsy procedure, but all reasonable efforts will be made to minimize pain. The biopsy procedure is done within the boundaries of the existing wound to avoid giving the patient a separate new wound. Bleeding is a possible complication, but the risk is low for the small biopsies and is reduced by using local anesthetics with epinephrine, and silver nitrate sticks are available in each room to cauterize biopsy sites as needed. Infection is also a potential risk; however, wound tissue biopsies are routinely performed as the standard of care in the CWC to diagnose wound infection. The biopsy site will be appropriately monitored for infection by the physician managing the wound during routine wound clinic visits.

The ABI test may result in temporary discomfort around the ankle or foot when the cuff is inflated, but does not present any further physical or medical risks. The wound fluid collection is non-invasive and does not present any risk. Study participants will not benefit directly from participation in this study. This research information has the potential of providing considerable benefits to wound care by identifying a key player that influences the closure of chronic diabetic wounds. Such knowledge should help develop novel biomarker and or miR-directed therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Willing and able to provide informed consent
* Willing and able to comply with protocol instructions, including all biopsies and study visits
* Diabetes Mellitus
* Chronic wounds (open >30d) of any etiology
* Subjects with Negative Pressure Wound Therapy (NPWT or also called a wound vac) (Note: Applies only to the miR-21 arm)

Exclusion Criteria:

* Revascularization surgery on the target wound within 60 days prior to enrollment
* Inadequate arterial supply, as evidenced by any of the following:
* Transcutaneous Oxygen Measurement (TcOM) < 30mmg
* Ankle Brachial Index (ABI) <0.7 or 1.3
* Toe Brachial Index (TBI) <0.6
* Subjects with marked immunodeficiency (HIV/AIDS, organ transplant patients and actively being treated for cancer)
* Trauma wounds
* Wounds closed or to be closed by flap or graft coverage
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 124 subjects with diabetic foot ulcers who have wound tissue oxygenation adequate to support wound healing
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Wound-edge endothelial miR-200b | 14 weeks
  This study aims to determine if elevated wound-edge endothelial miR-200b and attenuated wound macrophage miR-21 levels are barriers to wound healing (closure) in diabetic wounds.
Wound macrophage isolation to determine miR-21 | 14 weeks
  To determine if ex vivo supplementation of miR-21 mimic and recombinant MFG-E8 resolve inflammation in wound macrophages isolated from Negative Pressure Wound Therapy sponges from diabetic wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - OSU Hospital East, Columbus, Ohio
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio

REFERENCES:
- [Background] Chan YC, Khanna S, Roy S, Sen CK. miR-200b targets Ets-1 and is down-regulated by hypoxia to induce angiogenic response of endothelial cells. J Biol Chem. 2011 Jan 21;286(3):2047-56. doi: 10.1074/jbc.M110.158790. Epub 2010 Nov 16. PMID 21081489
- [Background] Chan YC, Roy S, Khanna S, Sen CK. Downregulation of endothelial microRNA-200b supports cutaneous wound angiogenesis by desilencing GATA binding protein 2 and vascular endothelial growth factor receptor 2. Arterioscler Thromb Vasc Biol. 2012 Jun;32(6):1372-82. doi: 10.1161/ATVBAHA.112.248583. Epub 2012 Apr 12. PMID 22499991
- [Background] Chin D, Boyle GM, Theile DR, Parsons PG, Coman WB. The human genome and gene expression profiling. J Plast Reconstr Aesthet Surg. 2006;59(9):902-11. doi: 10.1016/j.bjps.2006.01.008. Epub 2006 Mar 9. PMID 16920579
- [Background] Gardner SE, Frantz RA, Doebbeling BN. The validity of the clinical signs and symptoms used to identify localized chronic wound infection. Wound Repair Regen. 2001 May-Jun;9(3):178-86. doi: 10.1046/j.1524-475x.2001.00178.x. PMID 11472613
- [Background] Parsek MR, Singh PK. Bacterial biofilms: an emerging link to disease pathogenesis. Annu Rev Microbiol. 2003;57:677-701. doi: 10.1146/annurev.micro.57.030502.090720. PMID 14527295
- [Background] Roy S, Khanna S, Rink C, Biswas S, Sen CK. Characterization of the acute temporal changes in excisional murine cutaneous wound inflammation by screening of the wound-edge transcriptome. Physiol Genomics. 2008 Jul 15;34(2):162-84. doi: 10.1152/physiolgenomics.00045.2008. Epub 2008 May 6. PMID 18460641
- [Background] Roy S, Patel D, Khanna S, Gordillo GM, Biswas S, Friedman A, Sen CK. Transcriptome-wide analysis of blood vessels laser captured from human skin and chronic wound-edge tissue. Proc Natl Acad Sci U S A. 2007 Sep 4;104(36):14472-7. doi: 10.1073/pnas.0706793104. Epub 2007 Aug 29. PMID 17728400
- [Background] Schafer M, Werner S. Transcriptional control of wound repair. Annu Rev Cell Dev Biol. 2007;23:69-92. doi: 10.1146/annurev.cellbio.23.090506.123609. PMID 17474876
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Shilo S, Roy S, Khanna S, Sen CK. Evidence for the involvement of miRNA in redox regulated angiogenic response of human microvascular endothelial cells. Arterioscler Thromb Vasc Biol. 2008 Mar;28(3):471-7. doi: 10.1161/ATVBAHA.107.160655. Epub 2008 Feb 7. PMID 18258815
- [Background] Shilo S, Roy S, Khanna S, Sen CK. MicroRNA in cutaneous wound healing: a new paradigm. DNA Cell Biol. 2007 Apr;26(4):227-37. doi: 10.1089/dna.2006.0568. PMID 17465889
- [Background] Hopf HW, Ueno C, Aslam R, Burnand K, Fife C, Grant L, Holloway A, Iafrati MD, Mani R, Misare B, Rosen N, Shapshak D, Benjamin Slade J Jr, West J, Barbul A. Guidelines for the treatment of arterial insufficiency ulcers. Wound Repair Regen. 2006 Nov-Dec;14(6):693-710. doi: 10.1111/j.1524-475X.2006.00177.x. No abstract available. PMID 17199834
- [Background] Padberg FT, Back TL, Thompson PN, Hobson RW 2nd. Transcutaneous oxygen (TcPO2) estimates probability of healing in the ischemic extremity. J Surg Res. 1996 Feb 1;60(2):365-9. doi: 10.1006/jsre.1996.0059. PMID 8598670
- [Background] Wutschert R, Bounameaux H. Determination of amputation level in ischemic limbs. Reappraisal of the measurement of TcPo2. Diabetes Care. 1997 Aug;20(8):1315-8. doi: 10.2337/diacare.20.8.1315. PMID 9250461